CLINICAL TRIAL: NCT00234273
Title: Effects Rehabilitation Programme in Adapted Physical Activity (APA) Among Type 2 Diabetics Persons
Brief Title: APAD2: Effects of Rehabilitation Programme in Adapted Physical Activity (APA) Among Type 2 Diabetics
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recrutment
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DCIC 03 09
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: NIDDM
Keywords: Adapted Physical Activity; Quality of life; cardiovascular risk; teaching; Directly Observed Therapy; Physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Directly Observed Therapy; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic education combining dietary and rehabilitation (Experimental): Therapeutic education combining dietary and rehabilitation (APA)
  Interventions: Procedure: Rehabilitation programme in Adapted Physical Activity (APA); Behavioral: Therapeutic education primarily focused on dietary
- Therapeutic education primarily focused on dietary (Active Comparator): Therapeutic education primarily focused on dietary
  Interventions: Behavioral: Therapeutic education primarily focused on dietary

INTERVENTIONS:
Procedure: Rehabilitation programme in Adapted Physical Activity (APA)
  Arms: Therapeutic education combining dietary and rehabilitation
Behavioral: Therapeutic education primarily focused on dietary

SUMMARY:
The principal objective is to assess and analyze the effects of a six month programme in Adapted Physical Activity (APA) on physical activity, compliance, and insulin resistance among type 2 diabetics.

DETAILED DESCRIPTION:
Clinical trial with direct individual profit. Study phase 2. Study center: University Hospital Grenoble Principal investigator: Pr. Serge HALIMI Sponsor: University Hospital Grenoble

The principal objective is to assess and analyze the effects of a six month programme in Adapted Physical Activity (APA) on physical activity, compliance, and insulin resistance among type 2 diabetics.

Secondary objectives are to assess and analyze the effects of a six month programme in APA of:

* arterial tension
* weight, body composition and abdominal perimeter
* quality of life
* treatment dosage
* number of hospitalisation thick a diabetes complication acute for one year and for each patient Compare two exercise's intensity: first lactate threshold (SL1) and crossover (PCGL).

Inclusion criteria:

* type 2 diabetics
* age > 40 years
* first education in Education Diabetics Department of University Hospital Grenoble
* sedentary patients
* HbA1c > 7%-
* BMI > 25
* to be affiliate disease assurance
* to give consent written and inform

Judgment criteria for physical activity compliance:

* leisure time physical activity: Modifiable Activity Questionnaire
* training note-book

Judgment criteria for resistance insulin:

* Crossover (PCGL)
* HOMA and FIRI index
* HbA1c

Programme test: Rehabilitation programme in Adapted Physical Activity (APA)

Programme test period: 6 months

Study total period: 28 months

Study period for each patient: 18 months

Safety criteria: clinical compendium undesirable events

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetics
* Age > 40
* First education in the Education Diabetics Department of the University Hospital Grenoble
* Sedentary patients
* Hemoglobin A1c (HbA1c) > 7%
* Body mass index (BMI) > 25
* To be affiliated with disease assurance
* To give written and informed consent

Exclusion Criteria:

* Foot sore < six months
* Renal disease - proteinuria stage
* Contraindication for exercise
* VO2 max > 120% Wassermann standard
* Coronary pathology non-stabilization
* Arteriopathy stage 2 non-compensation
* Osteo-articular crippling problem
* Geographically distant

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Increase physical activity compliance long-term | 6 months after the beginning of the program
  Modifiable Activity Questionnaire (MAQ
Lessen insulin resistance | 6 months after the beginning of the program
  HOMA (Homeo-stasis model assessment), HbA1c, PCGL

SECONDARY OUTCOMES:
Improve the quality of life | 6 months after the beginning of the program
  Short Form-36 Health Survey Questionnary (SF-36)
Improve the arterial tension | 6 months after the beginning of the program
  arterial tension
Lessen the weight | 6 months after the beginning of the program
  weight

CONTACTS AND LOCATIONS:
Overall Officials: HALIMI Serge, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Halimi S. Therapeutic strategies for type 2 diabetes. Rev Prat HALIMI, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (4):
- France (4):
  - Department of Endocrinology, Diabetology and Nutrition, Grenoble, Auvergne-Rhône-Alpes
  - Endocrinology, Diabetology and Nutrition - University Hospital of Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Endocrinology, Diabetology and Nutrition Department - University Hospital of Grenoble, Grenoble
  - HALIMI Serge, Grenoble

REFERENCES:
- [Result] Bouvard S, Faure P, Roucard C, Favier A, Halimi S. Characterization of free radical defense system in high glucose cultured HeLa-tat cells: consequences for glucose-induced cytotoxicity. Free Radic Res. 2002 Sep;36(9):1017-22. doi: 10.1080/107156021000006671. PMID 12448827
- [Result] Halimi S, Wion-Barbot N, Lambert S, Benhamou P. [Self-monitoring of blood glucose in type 2 diabetic patients. What could we propose according to their treatment?]. Diabetes Metab. 2003 Apr;29(2 Pt 2):S26-30. French. PMID 12746623
- [Result] Halimi S. [Therapeutic strategies for type 2 diabetes]. Rev Prat. 2003 May 15;53(10):1079-85. French. PMID 12846028
- [Result] Halimi S. [Is a new therapeutic class justified in the treatment of type 2 diabetes?]. Ann Endocrinol (Paris). 2002 Apr;63(2 Pt 2):1S7-11. French. PMID 12037511
- [Result] Halimi S, Charpentier G, Grimaldi A, Grenier JL, Baut F, Germain B, Magnette J. Effect on compliance, acceptability of blood glucose self-monitoring and HbA(1c) of a self-monitoring system developed according to patient's wishes. The ACCORD study. Diabetes Metab. 2001 Dec;27(6):681-7. PMID 11852377
- See also: PubMed — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi